CLINICAL TRIAL: NCT01083745
Title: Assessment of Blood and Follicular Fluid Immune Cell Constitution in Patients Undergoing in Vitro Fertilization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Adrian Ellenbogen, Hillel Yaffe Medical Center, IVF Unit
Other Study IDs: 022-10
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- IVF patients - 1: Poor responders
- IVF patients - 2: Good responders

SUMMARY:
The etiology of infertility in the majority of patients with poor response to ovarian stimulation remains unknown. This study will investigate the role of immune cells (T cells, B cells, dendritic cells and NK cells), that constitute the immune system which normally fights infection and cancer. We, the investigators, have found that specialized NK cells that help with new blood vessel formation, are found in the fluid surrounding the egg during IVF, only in patients with good response to ovarian stimulation. We now wish to expand our studies and correlate our findings to ovarian blood flow , as measured by 3D ultrasound and to the presence of other cells in the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Age 27-43 years
* Diagnosis of infertility due to endometriosis, severe male factor, tubal occlusion.
* Patient undergoing IVF

Exclusion Criteria:

* Body mass index (BMI) > 38 kg/m2
* Abnormal uterine cavity as evidenced by sonohysterogram or hysterosalpingography
* Any current use of systemic steroid medication or any infertility treatment within 3 months of study enrollment.
* Any contraindication to being pregnant and carrying a pregnancy to term.
* Any ovarian or abdominal abnormality that may interfere with adequate TVS evaluation.
* Absence of one or two ovaries
* Clinically relevant systemic disease (e.g., Insulin-dependent diabetes, adrenal dysfunction, organic intracranial lesion, polycystic ovarian syndrome, hyperprolactinemia, or hypothalamic tumor) or serious illness (Neoplasia).
* History (within past 12 months) or current abuse of alcohol or drugs.
* Administration of any investigational drugs within three months prior to study enrollment.
* Any medical condition that may interfere with the absorption, distribution, metabolism or excretion of the study drugs, gastrointestinal diseases, mal absorption syndromes and liver dysfunction
* Unexplained gynecological bleeding.
* Ejaculated sperm is not sufficient for ICSI
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study.
* Abnormal COH screening blood done for both partners, including: prolactin, thyroid stimulating hormone, HIV serology, Hepatitis B and C serology, Rubella, group and screen and syphilis serology prior to participation in study.
* Unwillingness to give written informed consent. Previous entry into this study or simultaneous participation in another clinical trial.

Ages: 27 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: IVF clinic patients in tertiary care center
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel